CLINICAL TRIAL: NCT01616043
Title: Clinical Application of GLYADERM. A Multicentre, Prospective, Randomized Controlled, Comparative Trial of Glyaderm and Split Thickness Skin Graft Versus Split Thickness Skin Graft Alone in Full Thickness Skin Defects
Brief Title: Glyaderm Clinical Evaluation Multicenter Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: delay in recruitment, lack of additional funding
Sponsor: Euro Tissue Bank (Other)
Collaborators: Dutch Burns Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/363; B67020108965 (Other Grant/Funding Number: Belgian registration number: B67020108965)
Record Dates: First submitted 2012-05-29; First posted 2012-06-11 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Full-thickness Skin Loss Due to Burn, Unspecified Site
Keywords: scar quality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glyaderm + STSG (Experimental): All included patients in this arm will undergo full thickness removal of the burned skin or adequate debridement of all necrotic tissue. The wounds of the patients will be covered with glycerol preserved allografts for wound bed preparation. At the second operation, 5-7 days after the first operation, the allografts are removed. If the wound bed is not suitable for grafting, additional wound bed preparation with allografts is required until the wound bed is satisfactory. If the wound bed is suitable for grafting, the wounds of the patients are covered with Glyaderm®. After 6-8 days the wounds are finally covered with a thin STSG.
  Interventions: Procedure: Glyaderm
- STSG alone (Other): All included patients in this arm will undergo full thickness removal of the burned skin or adequate debridement of all necrotic tissue. The wounds of the patients will be covered with glycerol preserved allografts for wound bed preparation. At the second operation, 5-7 days after the first operation, the allografts are removed. If the wound bed is not suitable for grafting, additional wound bed preparation with allografts is required until the wound bed is satisfactory. If the wound bed is suitable for grafting, the wounds are immediately covered with a thin STSG.
  Interventions: Procedure: STSG

INTERVENTIONS:
Procedure: Glyaderm — acellular dermis
  Other Names: dermal substitute
  Arms: Glyaderm + STSG
Procedure: STSG — autologous split skin only
  Other Names: autologous skin graft
  Arms: STSG alone

SUMMARY:
The healing of full thickness skin defects treated with a split thickness skin graft (STSG) is frequently associated with excessive scarring and contraction. The psychological burden of poor cosmesis of these scarred regions as well as functional problems due to skin tightness and decreased joint mobility cause a very significant morbidity in these patients. Application of a dermal substitute underneath the split skin may improve the quality of the scar. Glyaderm is a dermal substitute derived from human skin and due to the elastin in this substitute it will contribute to a long term improvement of pliability and function and a better esthetic outcome.

The main objective is to evaluate the difference in scar quality, after skin restoration of full thickness defects treated with Glyaderm® and STSG versus STSG alone. Secondary objectives are: to evaluate the percentage of Glyaderm® take before application of autografts, to compare healing time and percentage of autograft survival and bacterial load in full thickness defects treated with Glyaderm® and STSG versus STSG alone, and to conduct a concurrent cost-effectiveness and health related quality of life study (i.e. cost utility analysis).

The study is an interventional, prospective, randomized and controlled interactive web based, study in a multicentre setting. Patients with full thickness burn wounds or full thickness skin defects will be evaluated before enrolment. A total of 120 patients will be included.

All included patients will undergo full thickness removal of the burned skin or adequate debridement of all necrotic tissue. The wounds of the patients will be covered with glycerol preserved allografts for wound bed preparation. At the second operation, 5-7 days after the first operation, the allografts are removed. If the wound bed is not suitable for grafting, additional wound bed preparation with allografts is required until the wound bed is satisfactory. If the wound bed is suitable for grafting, the patient is randomized to the Glyaderm® group or the control group. The wounds of the patients randomized to the Glyaderm® group are covered with Glyaderm®. After 6-8 days the wounds are finally covered with a thin STSG. In the control group, the wounds are immediately covered with a thin STSG.

Up to one year after complete wound closure, patients are followed-up for scar evaluation and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All clearly full thickness burns or skin defects (TBSA Full Thickness Burn < 30%) as clinically evaluated by two plastic surgeons and/or specialist burn surgeons
* Possibility to follow the complete treatment schedule until final graft take and subsequently wound healing and finally participation in the follow-up schedule
* Informed consent has been obtained.

Exclusion Criteria:

* All partial thickness burns that can heal by conservative treatment
* TBSA > 30 %
* Study wound < 100 cm² or > 800 cm²
* Age of the patient < 18 year
* No follow-up until wound closure or withdrawal before start of follow-up
* Patient has any condition(s) that seriously compromises the patient's ability to complete this study.
* Patient has participated in another study utilizing an investigational drug within the previous 30 days
* Patient has one or more medical condition(s), diabetes, including renal, hepatic, hematologic, neurologic, or immune disease that in the opinion of the investigator would make the patient an inappropriate candidate for this study
* No informed consent before start of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
scar quality | 12 months after wound closure
  The quality of the scar is measured with objective tools and subjective scar scacles. The elasticity of the scar is measured with the Cutometer® MPA 850 (Courage & Khazaka electronic GmbH) Adapted Vancouver Scar Scale, Patient and Observer Scar Assessment Scale, Ghent contour scale, Tewameter TM 300 for trans epidermal water loss, Corneometer CM 825 for hydration of the stratum corneum, Mexameter MX 18 for erythema and melanin, Reviscometer RVM 600 for the direction of collagen and elastin in the skin Finally a total score is defined.

SECONDARY OUTCOMES:
percentage of Glyaderm take | before autograft application (5-7 days after Glyaderm application)
  1. visual assessment of Glyaderm ingrowth

CONTACTS AND LOCATIONS:
Overall Officials: Ali Pirayesh, MD, Principal Investigator — UZ Gent, Belgium
Locations (6):
- Belgium (3):
  - Hospital Network Antwerp - site Stuivenberg, Antwerp
  - Militairy Hospital neder over heembeek, Brussels
  - Ghent University Hospital (B), Ghent
- General Hospital of Athens "G. Gennimatas" (GR), Athens, Greece
- Maasstad Ziekenhuis, Rotterdam, Netherlands
- Hospital Universitari Vall d'Hebron, Barcelona, Spain